CLINICAL TRIAL: NCT03300102
Title: A Single Site Study Accessing the Acceptability and Feasibility of Patient-specific 'Tumouroids' as Personalised Treatment Screening Tools
Brief Title: Acceptability and Feasibility Study of Patient-specific 'Tumouroids' as Personalised Treatment Screening Tools
Acronym: Tumouroids
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 17/0351
Record Dates: First submitted 2017-07-12; First posted 2017-10-03 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Cancer
Keywords: personalised medicine
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic; Tissue and Organ Procurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected or confirmed renal cell carcinoma: Patients with suspected or confirmed renal cell carcinoma who have consented will either donate tissue, or complete a structured questionnaire or a semi-structured interview. Not all patients will have all three interventions, each patient must have at least one.
  Interventions: Other: Questionnaires, interviews and or tissue donation

INTERVENTIONS:
Other: Questionnaires, interviews and or tissue donation — Subjects will be asked to complete either structured questionnaires, semi-structured interviews or donate tissue. There will be some overlap, but each subject does not have to do all three interventions.

SUMMARY:
In England, more than three hundred thousand people are diagnosed with cancer each year. The diagnostic and treatment pathways for multiple cancers have greatly developed over the past decade. However, novel treatments are expensive and currently discrimination between responders and non-responders is still suboptimal. There is a pressing need to develop tools that allow for better disease characterisation and stratification. Personalised medicine, whereby prevention, diagnosis, and treatment of diseases is aimed at the individual level, is a growing field. Predicting patient-specific treatment response is challenging as response depends not only on the characteristics of cancer cells but also on how these cells interact with their immediate surrounding environment and on how the tumour interacts with the host. A simplistic model is therefore insufficient to predict treatment response. Complex, patient-derived animal models have been used to this effect but are expensive, may take up to 6 months to provide clinically relevant answers, and pose ethical issues. In the past in vitro models lacked complexity as they were based solely on the two-dimensional (2D) growth of cancer cells. Nowadays the use of 3D tumour models has provided an extra level of complexity to in vitro studies. With these models it is possible to recreate tumour characteristics that were lost in 2D, such as cell-cell interaction between cancer cells and between cancer and stromal cells, cell-matrix interaction, or hypoxia.

The investigators have developed a 3D complex tumour model - named tumouroid. Using this model, preliminary work has been undertaken which allows the growth of patient-derived tumouroids using primary cancer cells from patients.

This personalised platform can be challenged by therapeutics used in clinical practice and response to treatment can be assessed via appropriate assays.

The study goals are twofold:

To assess patient acceptability to the use of patient derived tumour models for future decision-making, and To assess the feasibility of generating patient derived renal cancer tumouroids and using them as platforms to test drug response.

DETAILED DESCRIPTION:
This trial is a prospective tissue collection of renal cell carcinoma samples, including collection of data using both structured Likert 12 item questionnaires and semi structured interviews to assess acceptability. With the development of patient-derived tumouroids the investigators would like to overcome the current over-simplified strategies that focus on genetic markers as predictors of response. In the future, the investigators hope to establish tumouroids as a personalised platform to predict patient response to treatment that is more cost-efficient and poses less ethical issues than animal platforms.

This project will assess if patient-derived tumouroids can be therapeutically challenged and if patients would be willing to accept that such platform to guide clinical treatment decision making.

This study is designed to assess primarily patient acceptability. Acceptability will be elicited using Likert scale non-validated questionnaires and in a semi-structured interview in which the views and preferences relating the acceptability or otherwise of the patient derived tumour models and their impact on future decision making will be explored.

The study will also assess feasibility of building tumouroids and challenging them. Feasibility will address the successful transition between the critical phases of generating a viable and responsive tumour model. This begins with the extraction of cancer cells from the explanted tumour and ends with the determination of a response or otherwise to a therapeutic challenge of the viable tumour model at a range of in vitro concentrations.

The findings of this study will be presented at conference(s) and manuscripts will be submitted to appropriate journals for publication.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old), of either gender, able to provide consent;
* Suspected or confirmed renal cell carcinoma;
* Signed informed consent by patient

Exclusion Criteria:

* Non-English speaker;
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients aged 18 or over, sufficient command of English language to complete consent forms and questionnaires, suspected or confirmed renal cell carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Acceptability | Up to 10 weeks after consent
  Measured using a Likert scale non-validated structured questionnaire and/or complete a semi structured interview.

SECONDARY OUTCOMES:
Feasibility : Number of tumour tissue samples collected | Up to 10 weeks after consent
  Number of tumour tissue samples that can be collected within the time frame from consented patients this will be counted.
Feasibility : Gross morphology, weight and size of each sample | Up to 10 weeks after consent
  Each sample obtained will be weighed and measured.
Feasibility : Cell count after isolation | Up to 10 weeks after consent
  A physical count of the number of cells isolated from each sample will be collected.
Feasibility: Cell growth method and time | 10 days after tumouroid establishment
  Measurements will be taken of each tumouroid as it grows, each tumouroid will be given ten days to grow at day ten drug challenge will begin..
Feasibility: Drug concentrations tested | On day 10 after tumouroid establishment
  A log will be kept of the drug concentrations used on all tumouroids.
Feasibility: Duration of drug exposure | 5 days of drug exposure
  Number of days tumouroid was exposed to drug
Feasibility: Drug challenge response | within 6 days of the end of drug exposure.
  At the end of 5 days of drug exposure tumouroids will be assessed for response to the drug using a commercially available kit that assesses cell metabolism and viability. In addition, tumouroids will be fixed so that cell morphology will be assessed within 6 days of the end of drug exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Emberton, Principal Investigator — Professor of Interventional Oncology, UCL
Locations (2):
- United Kingdom (2):
  - Surgical & Interventional Trials Unit, London
  - Royal Free Hospital, London

REFERENCES:
- [Derived] Tran MGB, Neves JB, Stamati K, Redondo P, Cope A, Brew-Graves C, Williams NR, Grierson J, Cheema U, Loizidou M, Emberton M. Acceptability and feasibility study of patient-specific 'tumouroids' as personalised treatment screening tools: Protocol for prospective tissue and data collection of participants with confirmed or suspected renal cell carcinoma. Int J Surg Protoc. 2019 Apr 2;14:24-29. doi: 10.1016/j.isjp.2019.03.019. eCollection 2019. PMID 31851732